CLINICAL TRIAL: NCT05279235
Title: A Multi-center, Double-blinded, Randomized, Phase III Study to Evaluate the Efficacy and Safety of JT001 (VV116) Compared With Favipiravir in Participants With Moderate to Severe Coronavirus Disease 2019 (COVID-19)
Brief Title: Efficacy and Safety of JT001 (VV116) Compared With Favipiravir
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Development strategy adjustment
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JT001-006-III-COVID-19
Record Dates: First submitted 2022-03-08; First posted 2022-03-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-02

CONDITIONS: Moderate to Severe COVID-19
MeSH Terms: interventions — GS-621763; favipiravir

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JT001& Favipiravir Placebo (Experimental): JT001 (VV116):Day 1: 600mg, Q12H X 1 day; Day 2~5: 300mg, Q12H X 4 days Favipiravir placebo:Day 1: 1600mg, Q12H X 1 day; Day 2~5: 600mg, Q12H X 4 days
  Interventions: Drug: JT001; Drug: Favipiravir placebo
- Favipiravir & JT001 Placebo (Active Comparator): Favipiravir:Day 1: 1600mg, Q12H X 1 day; Day 2~5: 600mg, Q12H X 4 days JT001 (VV116) placebo:Day 1: 600mg, Q12H X 1 day; Day 2~5: 300mg, Q12H X 4 days
  Interventions: Drug: JT001 placebo; Drug: Favipiravir

INTERVENTIONS:
Drug: JT001 — Day 1: 600mg, Q12H X 1 day; Day 2~5: 300mg, Q12H X 4 days
  Other Names: VV116
  Arms: JT001& Favipiravir Placebo
Drug: JT001 placebo — Day 1: 600mg, Q12H X 1 day; Day 2~5: 300mg, Q12H X 4 days
  Other Names: VV116 placebo
  Arms: Favipiravir & JT001 Placebo
Drug: Favipiravir — Day 1: 1600mg, Q12H X 1 day; Day 2~5: 600mg, Q12H X 4 days
  Arms: Favipiravir & JT001 Placebo
Drug: Favipiravir placebo — Day 1: 1600mg, Q12H X 1 day; Day 2~5: 600mg, Q12H X 4 days
  Arms: JT001& Favipiravir Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JT001 (VV116) for the Treatment of Coronavirus Disease 2019 (COVID-19) in participants with moderate to severe COVID-19.

DETAILED DESCRIPTION:
Screening Interested participants will sign the appropriate informed consent form (ICF) prior to completion of any study procedures.

The investigator will review symptoms, risk factors and other non-invasive inclusion and exclusion criteria prior to any invasive procedures. If the participant is eligible after this review, then the site will perform the invasive procedures to confirm eligibility.

Treatment and Assessment Period

This is the general sequence of events during the 29-day treatment and assessment period:

* Complete baseline procedures and sample collection
* Participants are randomized to an intervention group
* Participants receive study intervention (Q12H X 5 days), and
* Complete all safety monitoring.
* Blood samples collection

ELIGIBILITY:
Inclusion Criteria:

1. Participants of 18 years of age or older, at the time of signing of informed consent
2. Participants who have a positive SARS-CoV-2 test result
3. Participants who have one or more COVID-19 symptoms, such as fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, shortness of breath with exertion
4. Participants who have SpO2≤93% on room air at sea level or PaO2/FiO2≤ 300
5. Participants who must agree to adhere to contraception restrictions
6. Participants who understand and agree to comply with planned study procedures
7. Participants or legally authorized representatives can give written informed consent approved by the Ethical Review Board governing the site
8. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Participants who are judged by the investigator as likely to progress to critical COVID-19 prior to randomization.
2. Participants who require mechanical ventilation or anticipated impending need for mechanical ventilation
3. Participants who are suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention
4. Participants who have eye disease (such as inflammation, Vessel deformity, retinal hemorrhage or decollement, optic nerve lesion, or fundus lesion)
5. Participants who have any of the following conditions when screening:

   * ALT or AST>1.5 ULN
   * Systolic blood pressure < 90 mm Hg
   * Diastolic blood pressure < 60 mm Hg
   * Requiring vasopressors
   * Multi-organ dysfunction/failure
6. Participants who have known allergies to any of the components used in the formulation of the interventions
7. Any medical condition, which in the opinion of the Investigator, will compromise the safety of the participant
8. Participants who have received a SARS-CoV-2 monoclonal antibody treatment or prevention, or antiviral treatment (including the investigational treatment)
9. Participants who have received convalescent COVID-19 plasma treatment
10. Participants who have received SARS-CoV-2 vaccine prior to randomization.
11. Participants who have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed
12. Participants who are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
13. Female who is pregnant or breast-feeding or plan to be pregnant within this study period
14. Male whose wife or partner plan to be pregnant within this study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
progression of COVID-19 | Up to 29 days
  Percentage of the participants who have progression of COVID-19, defined as progress to critical COVID-19* or death from any cause, through Day 29

SECONDARY OUTCOMES:
AEs and SAEs | Up to 29 days
  Safety assessments such as AEs and SAEs through Day 29
Progress, Death | Up to 29 days
  Percentage of participants who experience these events by Day 29
  * Progress to critical COVID-19
  * Death from any cause
WHO 11-point ordinal outcome scale | Day 3, 5, 7, 10 and 29
  The change of WHO 11-point ordinal outcome scale from baseline to Day 3, 5, 7, 10 and 29(0-uninfected,10-dead)
The change of Chest CT scan | Day 7 and 10
  The change of Chest CT scan from baseline to Day 7 and 10（Percentage of lung involved）
SARS-CoV-2 clearance | Day 3, 5 ,7 and 10
  Percentage of participants achieve SARS-CoV-2 clearance at Day 3, 5 ,7 and 10

OTHER OUTCOMES:
SARS-CoV-2 viral genetic variation | Day 1
  SARS-CoV-2 viral genetic variation

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ma, Master, Study Director — Shanghai Junshi Bioscience Co., Ltd.
Locations (2):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China
- Specialized lnfectious Diseases Hospital No2 of Zangiota District, Tashkent, Tashkent Region, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided